CLINICAL TRIAL: NCT05785494
Title: Web-based Support to Promote Preparedness for Caregiving Among Family Caregivers of Patients With Advanced Cancer
Brief Title: Web-based Support for Family Caregivers of Patients With Advanced Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ersta Sköndal University College (Other)
Responsible Party: Principal Investigator, Anette Alvariza, Professor, Ersta Sköndal University College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MarieCederschiöldUniversity
Record Dates: First submitted 2023-02-27; First posted 2023-03-27 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Family; End of Life; Cancer Metastatic; Chronic Illness
Keywords: Palliative care; Family caregiver; Web-based support; Intervention
MeSH Terms: conditions — Death; Neoplasm Metastasis; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Access to web-site
  Interventions: Other: Narstaende.se
- Control (No Intervention): Standard care

INTERVENTIONS:
Other: Narstaende.se — Web-site with supportive information, videos and chat forum targeting family caregivers of patients with life-threatening illness.
  Arms: Intervention

SUMMARY:
For family caregivers of patients with advanced cancer, preparedness for caregiving is crucial for maintaining health and quality of life both during care and after the death of the patient. This project contributes to earlier research funded by the Swedish Cancer Society, about an intervention that was delivered by a multi-professional team and proved to be successful in promoting preparedness. However, such interventions are often costly and logistically challenging. In addition, the Covid-19 pandemic has further significantly raised the need for digital alternatives in healthcare. As a possible solution, an evidence-based intervention, narstaende.se, has been developed consisting of recorded videos of conversations between clinicians and family caregivers (actors), linked to informational texts and a moderated chat forum. The intervention was pilot tested during 2020 and 2021, exploring feasibility, content and family caregivers' experiences. As preliminary results are promising, the intervention is taken one step further and tested as a web-based intervention in a larger scale.

ELIGIBILITY:
Inclusion Criteria:

* Being a family caregiver, over 18 years of age, to a person with life-threatening illness cared for in specialized home care.

Exclusion Criteria:

* Not being able to communicate in Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Preparedness for caregiving | At baseline (before intervention), change from baseline after 4-6 weeks (follow-up 1) and after 8-10 weeks (follow-up 2)
  Preparedness for caregiving scale (PCS)

SECONDARY OUTCOMES:
Change in Quality of Life | At baseline (before intervention), change from baseline after 4-6 weeks (follow-up 1) and after 8-10 weeks (follow-up 2)
  The Quality of Life in Life-Threatening Illness Family caregiver version (QOLLTI-F)
Change in health | At baseline (before intervention), change from baseline after 4-6 weeks (follow-up 1) and after 8-10 weeks (follow-up 2)
  RAND- 36
Change in Anxiety and Depression | At baseline (before intervention), change from baseline after 4-6 weeks (follow-up 1) and after 8-10 weeks (follow-up 2)
  The Hospital Anxiety and Depression Scale (HADS)
Change in pre-loss grief | At baseline (before intervention), change from baseline after 4-6 weeks (follow-up 1) and after 8-10 weeks (follow-up 2)
  Prolonged Grief-12
Change in post-loss grief | At baseline (before intervention), change from baseline after 4-6 weeks (follow-up 1) and after 8-10 weeks (follow-up 2)
  Prolonged Grief-13

CONTACTS AND LOCATIONS:
Locations (1):
- Marie Cederschiöld University, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bauman C, Wallin V, Doveson S, Furst P, Hudson P, Kreicbergs U, Alvariza A. The family caregiver-targeted web-based intervention "narstaende.se" facilitated everyday life for couples facing life-threatening illness: A qualitative study. Palliat Med. 2025 May;39(5):574-583. doi: 10.1177/02692163251327893. Epub 2025 Apr 12. PMID 40219770